CLINICAL TRIAL: NCT03661593
Title: Aniseikonia in Epiretinal Membranes
Brief Title: Aniseikonia in Epiretinal Membrane Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Glostrup University Hospital, Copenhagen (Other)
Responsible Party: Principal Investigator, Therese Krarup, Principal investigator, Glostrup University Hospital, Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: H-16020057
Record Dates: First submitted 2018-08-31; First posted 2018-09-07 (Actual); Last update posted 2018-09-07 (Actual); Status verified 2018-09

CONDITIONS: Epiretinal Membrane
MeSH Terms: conditions — Epiretinal Membrane

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Masking done by a third person following computer randomization
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cataract guideline (Experimental): In this patients we follow cataract guideline and correct the patients ametropia during the cataract surgery
  Interventions: Other: Cataract guideline
- Standard refraction (No Intervention): The patients gets an IOL ensuring his preoperatively refraction

INTERVENTIONS:
Other: Cataract guideline — The patients gets an IOL according to cataract guideline correcting the ametropia
  Arms: Cataract guideline

SUMMARY:
Examination of aniseikonia in epiretinal membranes patients before and after surgery

DETAILED DESCRIPTION:
Phakic patients woth epiretinal membranes are examined for aniseikonia and refractive status before and after surgery. Follow up is one year.

ELIGIBILITY:
Inclusion Criteria:

* Epiretinal membrane Phakic on both eyes

Exclusion Criteria:

* no previous eye surgeries
* refractive status +/- 2 seq

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-01 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Aniseikonia | 1 year
  Measure amount of aniseikonia by measuring aniseikonia with both computer program aniseikonia inspector and the New Aniseikonia test

CONTACTS AND LOCATIONS:
Locations (1):
- Eye department, Nordre ringvej 56, Copenhagen, Glostrup, Denmark

IPD SHARING:
Plan to Share IPD: No
No planing on sharing